### **Short Title:**

# Statistical Analysis Plan CLY935-C013 / NCT04476784

**Full Title:** 

# Statistical Analysis Plan CLY935-C013

| Replacement Soft Silicone Hydrogel Contact Len | <b>Protocol Title:</b> | Clinical Assessment of a Daily Wear Monthly |
|---|---|---|
| | | Replacement Soft Silicone Hydrogel Contact Lens |
| Approvals: See last page for electronic approvals | Approvals: | See last page for electronic approvals |
| Job Notes: | Job Notes: | |
| This | | This |

version of the Statistical Analysis Plan is based on Version 1.0 of the study protocol.

Document ID: V-CLN-0000838

Status: Approved, Version: 2.0 Approved Date: 02 Dec 2020 Page 2 of 16

### **Executive Summary:**

Key Objective:

The primary objective of this study is to evaluate visual acuity (VA) of the investigational Phoenix contact lens.

Decision Criteria for Study Success:

Decision criteria for study success are not applicable for this study.

## **Table of Contents**

| Statistic | cal Analysis Plan CLY935-C013 | 1 |
|-----------|-----------------------------------------------------|----|
| Table of | f Contents | 3 |
| List of T | Tables | 4 |
| 1 | Study Objectives and Design | 5 |
| 1.1 | Study Objectives | 5 |
| 1.2 | Study Description | 5 |
| 1.3 | Randomization | 6 |
| 1.4 | Masking | 6 |
| 2 | Analysis Sets | 6 |
| 2.1 | Safety Analysis Set | |
| 2.2 | Full Analysis Set. | |
| 3 | Subject Characteristics and Study Conduct Summaries | 7 |
| 4 | Effectiveness Analysis Strategy | 7 |
| 4.1 | Effectiveness Endpoints | 8 |
| 4.2 | Effectiveness Hypotheses | 9 |
| 4.3 | Statistical Methods for Effectiveness Analyses | 9 |
| 5 | Safety Analysis Strategy | 11 |
| 5.1 | Safety Endpoints | 11 |
| 5.2 | Safety Hypotheses | 12 |
| 5.3 | Statistical Methods for Safety Analyses | 12 |
| 5.3.1 | Adverse Events | |
| 5.3.2 | Biomicroscopy Findings/Slit Lamp Examination | 13 |

Page 4 of 16

Status: Approved, Version: 2.0 Approved Date: 02 Dec 2020

| 5.3.3 | Device Deficiencies | 13 |
|------------|------------------------------------|----|
| 7 | Sample Size and Power Calculations | 14 |
| 8 | References. | 14 |
| 9 | Revision History | 14 |
| 10 | Appendix | 15 |
| | List of Tables | |
| Table 1-1 | Study Description Summary | 5 |
| Table 10-1 | | |

## 1 Study Objectives and Design

## 1.1 Study Objectives

#### PRIMARY OBJECTIVE

The primary objective of this study is to evaluate distance VA of the investigational Phoenix contact lens.



# 1.2 Study Description

Key components of the study are summarized in Table 1-1.

Table 1-1 Study Description Summary

| Study Design | Prospective, randomized, bilateral crossover, double-masked |
|---|---|
| Study Population | Volunteer subjects aged 18 years or older who are current |
| | wearers of spherical weekly/monthly soft contact lenses in both |
| | eyes with at least 3 months wearing experience, with a |
| | minimum wearing time of 5 days per week and 10 hours per |
| | day. |
| | Planned to enroll: ~65 |
| | Target to complete: 58 |
| Number of Sites | ~5 (US) |
| Test Product | (LID018869) |
| Control Product | CooperVision® Biofinity® contact lenses (Biofinity) |
| Planned Duration of | ~60 days total duration |
| Exposure | Test Product: ~30 days |
| | Control Product: ~30 days |
| Visits | Visit 1: Screen/Baseline/Dispense Pair 1 (Day 1) |
| | Visit 2: Day 30 Follow-up Pair 1 (Day 30 ±2 days) |
| | Visit 3: Dispense Pair 2 |
| | Visit 4: Day 30 Follow-up Pair 2/Exit (Day 30 ±2 days) |

#### 1.3 Randomization

A member of the Randomization Programming group at Alcon who is not part of the study team will generate the randomized allocation schedule(s) for lens sequence assignment. Randomization will be implemented in the Electronic Data Capture (EDC)/randomization integration system.

Subjects will be randomized in a 1:1 ratio to receive treatment in a crossover sequence of Test product then Control product or Control product then Test product, respectively.

#### 1.4 Masking

This study is double-masked.

### 2 Analysis Sets

### 2.1 Safety Analysis Set

Safety analyses will be conducted using the safety analysis set on a treatment-emergent basis. As such, the safety analysis set will include all subjects/eyes exposed to any study lenses evaluated in this study. For treatment-emergent safety analyses, subjects/eyes will be categorized under the actual study lenses exposed in the corresponding lens sequence.

Adverse events occurring from the time of informed consent but prior to first exposure to study lenses will be summarized in subject listings.

# **2.2** Full Analysis Set

The full analysis set (FAS) is the set of all randomized subjects who are exposed to any study lenses evaluated in this study.



## 3 Subject Characteristics and Study Conduct Summaries

The following tables will be presented:

- Subject Disposition by Lens Sequence
- Analysis Sets by Lens
- Analysis Sets by Lens Sequence
- Subject Accounting by Lens Sequence
- Demographics Characteristics by Lens Sequence
- Baseline Characteristics by Lens Sequence



### 4 Effectiveness Analysis Strategy



All data obtained in evaluable subjects/eyes will be included in the analysis. No imputation for missing values will be carried out.

# 4.1 Effectiveness Endpoints

### **Primary Endpoint**

The primary endpoint is distance VA with study lenses, collected for each eye in logMAR.



# 4.2 Effectiveness Hypotheses

### **Primary Effectiveness**

No inferences are to be made on the primary effectiveness endpoint; therefore, no hypotheses are formulated.



### 4.3 Statistical Methods for Effectiveness Analyses

# 4.3.1 Primary Effectiveness Analyses

Descriptive statistics used for continuous variables will be presented.







# 5 Safety Analysis Strategy

# **5.1** Safety Endpoints

The safety endpoints are:

- Adverse events (AE)
- Biomicroscopy Findings/Slit Lamp Examinations

- Limbal hyperemia
- Bulbar hyperemia
- Corneal staining
- Conjunctival staining
- Palpebral conjunctival observations
- Corneal epithelial edema
- o Corneal stromal edema
- Corneal vascularization
- Conjunctival compression/indention
- Chemosis
- Corneal infiltrates
- Other findings
- Device deficiencies

#### 5.2 Safety Hypotheses

There are no formal safety hypotheses in this study. The focus of the safety analysis will be a comprehensive descriptive assessment of safety endpoints listed in Section 5.1.

#### 5.3 Statistical Methods for Safety Analyses

The analysis set for all safety analyses is the safety analysis set as defined in Section 2.1. Baseline will be defined as the last measurement prior to exposure to study lenses. For biomicroscopy data, baseline will be defined as Visit 1 for Period 1 and Visit 3 for Period 2. Safety variables will be summarized descriptively.

#### 5.3.1 Adverse Events

The applicable definition of an AE is in the study protocol. All AEs occurring from when a subject signs informed consent to when a subject exits the study will be accounted for in the reporting.



The following tables and supportive listings will be provided:

- Incidence of All Ocular Treatment-Emergent Adverse Events
- Incidence of Ocular Serious Treatment-Emergent Adverse Events
- Incidence of Ocular Significant Non-serious Treatment-Emergent Adverse Events
- Incidence of All Nonocular Treatment-Emergent Adverse Events
- Incidence of Nonocular Serious Treatment-Emergent Adverse Events
- Listing of All Ocular Treatment-Emergent Adverse Events
- Listing of All Nonocular Treatment-Emergent Adverse Events
- Listing of All Ocular Pre-Treatment Adverse Events
- Listing of All Nonocular Pre-Treatment Adverse Events



#### **5.3.3** Device Deficiencies

The following tables and supportive listings will be provided:

- Frequency of Treatment-Emergent Device Deficiencies
- Listing of Treatment-Emergent Device Deficiencies
- Listing of Device Deficiencies Prior To Treatment Exposure.



## **8** References

Not applicable.

# 10 Appendix

| Procedure / Assessment Procedure / Assessment Procedure / Assessment Procedure / Assessment Procedure / Assessment Pair 1 [Day 30 (± 2 days)] Informed Consent Demographics X Medical History X X X X X X X X X X X X X |
|---|
| Procedure / Baseline/ Dispense Pair 1 [Day 30 (± 2 days)] Informed Consent X Demographics X Medical History X X X X X X X X X X X X X |
| Demographics X Medical History X X X X Concomitant Medications X X X X |
| Medical History X X X X X X Concomitant Medications X X X X X X X |
| Concomitant X X X X X X |
| Medications X X X X X |
| Inclusion/Exclusion X |
| Habitual lens (brand, power*,care) |
| VA w/ habitual contact lens correction (OD, OS, Snellen distance) * |

| Randomization# | X | | | | |
|-----------------------------------------------------|---|---|---|---|-----|
| Dispense study lenses# | Х | | х | | (X) |
| VA w/ study lenses,<br>(OD, OS, logMAR<br>distance) | х | х | х | х | (X) |

| | LENS F | PAIR 1 | LENS P | AIR 2 | |
|---|---|---|---|---|---|
| Procedure /<br>Assessment | Visit 1<br>Screen/<br>Baseline/<br>Dispense<br>Pair 1<br>[Day 1] | Visit 2<br>Day 30<br>Follow-up<br>Pair 1<br>[Day 30<br>(± 2 days)] | Visit 3 Dispense Pair 2 [Day 1 after Washout] | Visit 4 Day 30 Follow-up Pair 2/Exit^ [Day30 (± 2 days)] | Unscheduled<br>visit |



| (* *) | (* 4) | (**) | <br>(**) |
|-------|-------|------|----------|

# Signature Page for V-CLN-0000838 v2.0



Signature Page for V-CLN-0000838 v2.0